CLINICAL TRIAL: NCT02264535
Title: A Pilot Study for Ginkgolides Meglumine Injection Skin Testing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Z-YXPU-ZS-IV4
Record Dates: First submitted 2014-09-04; First posted 2014-10-15 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-04

CONDITIONS: Allergy
Keywords: Allergy; Skin test; Ginkgolides Meglumine Injection
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.1mg/ml Ginkgolides Meglumine Injection (Experimental): Injection, 0.1mg/ml.
  Interventions: Drug: 0.1mg/ml Ginkgolides Meglumine Injection
- 1mg/ml Ginkgolides Meglumine Injection (Experimental): Injection, 1mg/ml.
  Interventions: Drug: 1mg/ml Ginkgolides Meglumine Injection
- 5mg/ml Ginkgolides Meglumine Injection (Experimental): Injection, 5mg/ml.
  Interventions: Drug: 5mg/ml Ginkgolides Meglumine Injection

INTERVENTIONS:
Drug: 0.1mg/ml Ginkgolides Meglumine Injection
  Arms: 0.1mg/ml Ginkgolides Meglumine Injection
Drug: 1mg/ml Ginkgolides Meglumine Injection
  Arms: 1mg/ml Ginkgolides Meglumine Injection
Drug: 5mg/ml Ginkgolides Meglumine Injection
  Arms: 5mg/ml Ginkgolides Meglumine Injection

SUMMARY:
This pilot study is designed to explore the optimal concentration and method of Ginkgolides Meglumine Injection skin testing and to evaluate the value of skin test in predicting any possible allergic reactions to Ginkgolides Meglumine Injection.

DETAILED DESCRIPTION:
Subjects will be enrolled in one of three groups with different doses to receive skin prick testing. Then they may be arranged to receive intradermal, subcutaneous injection or intravenous tests with different doses.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between the ages of 18 and 70(inclusive)at the time of signing the Informed Consent Form （ICF）.
* Subjects meet any one of the following requirements

  * No history of using any dugs containing bilobalide, Ginkgolide A, Ginkgolide B, Ginkgolide K (including Ginkgolides Meglumine Injection).
  * History of using any dugs containing bilobalide, Ginkgolide A, Ginkgolide B, Ginkgolide K (including Ginkgolides Meglumine Injection), and no allergy.
  * History of allergy to any dugs contain bilobalide, Ginkgolide A, Ginkgolide B, Ginkgolide K (including Ginkgolides Meglumine Injection).
  * History of allergy to any other drugs.
* Willingness to participate in the study as evidenced by signing the informed consent form.

Exclusion Criteria:

* Women in breastfeeding,menstrual or pregnancy period.
* Subjects are in the infectious disease, eczema, dermatitis, trauma,etc.
* Subjects meet any one of the following conditions

  * Used β-blockers within 2 days prior to starting this study.
  * Used H1 anti-histamines, imipramine, phenothiazine, Beta adrenaline etc. within 1 week prior to starting this study.
  * Used short-acting glucocorticoids drugs within 1 week prior to starting this study.
  * Topical used glucocorticoids drugs within 2 weeks prior to starting this study.
  * Used long-acting glucocorticoids drugs within 4 weeks prior to starting this study
* Subjects are currently participating or have participated in any other clinical trials within the prior 1 month of signing the ICF.
* Subjects have a history of allergic shock.
* Subjects who are not suitable for this clinical trial at the discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The rate of allergic reaction and analyze all kinds of positive reactions after skin prick test with different doses of Ginkgolides Meglumine Injection. | 15-20 minutes after skin prick tests.
The rate of allergic reaction and analyze all kinds of positive reactions after using intradermal tests of different doses of Ginkgolides Meglumine Injection. | 15-20 minutes after intradermal tests.

SECONDARY OUTCOMES:
The specificity and sensitivity with the different doses. | 15-20 minutes after prick-puncture and intradermal tests, 72 hours after subcutaneous test.
  Specificity (SPC) =TN/ (FP+TN); Sensitivity=TP/ (TP+FN). TP (true positive); TN (true negative); FP (false positive); FN (false negative). TP(true positive); TN(true negative); FP(false positive); FN(false negative).
Safety assessment will be based on adverse event reports, electrocardiogram, physical examinations and clinical laboratory tests. | within 7days before using Ginkgolides Meglumine Injectionand 3-10 days after using it.
  Only the participants who are allergic to the main components of Ginkgolides Meglumine Injection will be assessed in 3-10 days after using it by the investigators..

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Huang, Principal Investigator — Second Affiliated Hospital of Tianjin University of TCM
Locations (1):
- Second Affiliated Hospital of Tianjin University of TCM, Tianjin, China